CLINICAL TRIAL: NCT02449330
Title: Clinical Study for the Effect of Teneligliptin on the Left Ventricular Diastolic Dysfunction in Patients With Type 2 Diabetes Mellitus
Brief Title: Teneligliptin on the Progressive Left Ventricular Diastolic Dysfunction With Type 2 Diabetes Mellitus Study
Acronym: TOPLEVEL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Responsible Party: Principal Investigator, Masafumi Kitakaze, Director, National Cerebral and Cardiovascular Center, Japan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M26-43
Record Dates: First submitted 2015-05-17; First posted 2015-05-20 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- Teneligliptin in the inhibition test (Experimental): Patients showing E/e' by echocardiography less than 8 at base line and assigned as Teneligliptin treatment by randomization
  Interventions: Drug: Teneligliptin
- Other agents in the inhibition test (No Intervention): Patients showing E/e' by echocardiography less than 8 at base line and assigned as anti-diabetic agents except for DPP-4 inhibitors treatment by randomization
- Teneligliptin in the improvement test (Experimental): Patients showing E/e' by echocardiography more than 8 at base line and assigned as Teneligliptin treatment by randomization
  Interventions: Drug: Teneligliptin
- Other agents in the improvement test (No Intervention): Patients showing E/e' by echocardiography more than 8 at base line and assigned as anti-diabetic agents except for DPP-4 inhibitors treatment by randomization

INTERVENTIONS:
Drug: Teneligliptin
  Arms: Teneligliptin in the improvement test; Teneligliptin in the inhibition test

SUMMARY:
This is the clinical trial designed to assess the cardiac diastolic function of long term treatment with teneligliptin compared to that without teneligliptin in patients with type 2 diabetes mellitus by two arms; one includes patients showing E/e' by echocardiography less than 8, the other includes patients showing E/e' by echocardiography more than 8.

ELIGIBILITY:
Inclusion Criteria:

* Asians aged from 20 to 85 years old at baseline
* Patients with type 2 diabetes mellitus and including either A) or B) criteria.

A) Patients necessary to start the treatment using anti-diabetic agent(s) or to change the anti-diabetic agent(s).

B) Patients possible to change the anti-diabetic agent(s).

* Patients with left ventricular ejection fraction more than 40%
* Patients with written informed consent

Exclusion Criteria:

* Patients with type 1 diabetes mellitus
* Patients with slowly progressive type 1 diabetes mellitus positive for pancreatic islets related autoimmune antibody as GAD antibody or IA-2 antibody or ICA antibody
* Patients with diabetes mellitus caused by evident genetic factors
* Patients with diabetes mellitus caused by secondary factors as endocrine disease or liver disease
* Patients with diabetic ketoacidosis or hyperosmolar hyperglycemic syndrome
* Patients with any severe infectious diseases or planed any surgical treatments or suffered any severe traumas
* Patients with severe liver dysfunction
* Patients with hypophyseoprivic or adrenal insufficiency
* Patients under malnutrition or starved state or irregular caloric intake or calorie insufficiency or hyposthenia
* Patients judged to be unsuitable for the study as they are planning to exercise intensively
* Patients judged to be unsuitable for the study as they may drink excessively or abuse drugs
* Patients showing QT prolongation in the electrocardiogram
* Patients with any past histories of heart failure showing NYHA classification grade more than 3 at baseline
* Patients with any past histories of acute coronary syndrome or coronary intervention or cardiac surgery developed within 6 months
* Patients with any surgical past histories of mitral valve replacement or mitral valve repair or severe calcification of mitral valve
* Patients already treated with Teneligliptin
* Women with breast-feeding
* Pregnant women or patients who have possibilities of pregnancy
* Patients expected to live less than 3 years
* Patients with any past histories of drug hypersensitivity against Teneligliptin
* Patients already involved in any other interventional clinical trials or planned to be involved
* Patients judged to be inappropriate for the study by the doctors in charge

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 936 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change of the ratio of peak velocity of early transmitral diastolic filling by echocardiography (E) to early diastolic mitral annular velocity by tissue Doppler echocardiography (E/e') | Up to 2 years

SECONDARY OUTCOMES:
Total number of all-cause death | Up to 2 years
Total number of deaths by cardiovascular events | Up to 2 years
Total number of all-cause hospitalization | Up to 2 years
Total number of hospitalization by cardiovascular events | Up to 2 years
Total number of hospitalization by progression of heart failure | Up to 2 years
Total number of incidents for the addition or increase of the agents for heart failure by progression of heart failure | Up to 2 years
Change of the ratio of peak velocity of early transmitral diastolic filling (E) to late diastolic filling due to atrial contraction (E/A) by echocardiography | Up to 2 years
Change of the deceleration time (DT) by echocardiography | Up to 2 years
Change of the left atrium volume (LAV) by echocardiography | Up to 2 years
Change of the left ventricular end-diastolic diameter (LVDd), left ventricular end-systolic diameter (LVDs) and fractional shortening (%FS) by echocardiography | Up to 2 years
Change of the left ventricular mass index (LVMI) by echocardiography | Up to 2 years
Change of NYHA functional class | Up to 2 years
Change of plasma levels of NT-proBNP | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Cerebral and Cardiovascular Center, Suita, Japan